CLINICAL TRIAL: NCT07331662
Title: Comparative Effects of Intercostal and Thoracic Cage Stretching on Chest Expansion, Dyspnea, Oxygen Saturation in Asthma Patients
Brief Title: Intercostal and Thoracic Cage Stretching on Chest Expansion , Dyspnea ,Oxygen Saturation in Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S24C14G36006
Record Dates: First submitted 2025-12-29; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Asthma; Asthma (Diagnosis)
MeSH Terms: conditions — Asthma; Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intercostal stretching (Experimental): initially all patients will receive hotpack for 10-15 min then intercostal stretching will performed by them
  Interventions: Other: intercostal stretching
- Thoracic cage stretching (Experimental): initially all patients will receive hotpack for 10-15 min then intercostal stretching will performed by them
  Interventions: Other: thoracic cage stretching

INTERVENTIONS:
Other: thoracic cage stretching — thoracic cage stretching involve Sessions 4 times per week ,Intensity Stretch to the point of mild discomfort, but not pain. The goal is to feel a gentle stretch in the muscles being targeted, promoting flexibility without risking injury. Duration of Sessions: Each session should last about 30-40 minutes. Exercise Duration: Each exercise should involve 10repetitions ,Hold stretch for 10-30 sec. sets: 1-2, Rest for 1- 2 minutes between these two exercises. Types :chest opener stretch and overhead arm chest stretch
  Arms: Thoracic cage stretching
Other: intercostal stretching — intercostal stretching involve Sessions 4 times per week ,Intensity Stretch to the point of mild discomfort, but not pain. The goal is to feel a gentle stretch in the muscles being targeted, promoting flexibility without risking injury. Duration of Sessions: Each session should last about 30-40 minutes. Exercise Duration: Each exercise should involve 10repetitions ,Hold stretch for 10-30 sec. sets: 1-2, Rest for 1- 2 minutes between these two exercises. Types :lateral side bend stretch and torso rotational stretch
  Arms: intercostal stretching

SUMMARY:
The rationale of this study is to clarify distinct role of these two stretching techniques in pulmonary rehabilitation. Insight gained from this research could provide evidence based recommendations for implementing these therapeutic approaches, aiming to optimize symptoms in asthma patients. so improved respiratory function and muscular flexibility can empower individuals with asthma to better manage their condition, weakening of muscles, airflow obstruction , reduce the effort required for daily activities and engage more fully in physical and everyday tasks thereby enhancing overall quality of life.

DETAILED DESCRIPTION:
Asthma is a chronic respiratory disorder characterized by the inflammation and constriction of the airways, resulting in recurrent episodes of wheezing, shortness of breath, chest tightness, and coughing. This condition often results in the weakening and atrophy of muscles, particularly the key areas impacted include the respiratory muscles like intercostal muscles, muscles in the chest, shoulders, thoracic become weaker due to decreased physical activity. Stretching exercises can offer several benefits for individuals with asthma by improving overall lung function, enhancing muscle strength, and promoting relaxation. The objective of this study will be to evaluate the effects of intercostal and thoracic cage stretching on chest expansion, dyspnea, and oxygen saturation in asthma patients.

This study will be conducted as a randomized clinical trial with enrollment of 56 participants, that will divided equally into two groups. Group A will receive intercostal muscle stretching like lateral side bending stretch, torso rotational stretch, (4x\week) or Group B will undergo thoracic cage stretching like overhead arm chest stretch, chest opener stretch,(4x\week) .Study will be conducted for four weeks at sheikh zaid hospital Lahore, involving asthma patients both male and female. Key outcome measures will include chest expansion assessed using tape measure, dyspnea via Borg category scale, oxygen saturation via pulse oximeter. The non-probability convenient sampling technique, followed by random allocation using a lottery method ensure diverse yet unbiased sample. Pre, Post values will be noted. Data will be entered and analyzed by SPSS version 25 after checking normality of the data. Parametric and non-parametric test will be applied. Statistical significance will be set at P=0.05.

ELIGIBILITY:
Inclusion Criteria: Both males and females ,Diagnosed asthma patients ,All patients must have variable respiratory symptoms (cough, wheeze, shortness of breath, and/or chest tightness),All patients have to be clinically stable (ie, no exacerbations or changes in medication for the last 4 weeks before enrollment, sedentary life (doing <60 min of physical activity per week)

Exclusion Criteria: Other respiratory disease , Any orthopedic limitations ,Pediatric population ,Uncontrolled diabetes, hypertension ,Cardiovascular condition, pregnancy ,Smokers/ex-smokers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2025-04-17 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2025-12-17 (Actual)

PRIMARY OUTCOMES:
chest expansion | 4 week
  To measure chest expansion, we used a plastic tape measure. Stand straight with your arms relaxed at your sides, ideally wearing minimal clothing. First, measure your chest at rest by wrapping the tape around the widest part, under the armpits, across the nipples and at the level of xiphoid process, ensuring it's snug but not tight. Take this measurement after a normal exhalation. Next, for maximum expansion, take a deep breath and fully expand your chest, then measure again in the same spot at full inhalation. To find your chest expansion, subtract the resting measurement from the expanded measurement. It's best to repeat the process for accuracy,

SECONDARY OUTCOMES:
dyspnea | for 4 weeks
  The Borg Category Scale for dyspnea is a valuable tool for assessing breathlessness in asthma patients, ranging from 0 to 10, where 0 indicates no breathlessness and 10 represents maximal breathlessness. This scale enables patients to communicate their level of discomfort during various activities. During the study, participants were asked to rate their dyspnea before and after performing the exercises, providing a clear indication of any changes in their respiratory comfort. So we gained comprehensive insights into the effectiveness of the interventions in asthma patients.

OTHER OUTCOMES:
oxygen saturation | 4 week
  A pulse oximeter is a device that measures the oxygen saturation level in the blood (SpO₂) and the pulse rate. It works by emitting light through a person's fingertip or earlobe, analyzing how much light is absorbed by oxygenated and deoxygenated blood, and then estimating the blood's oxygen percentage.In this study for oxygen saturation we measured readings pre and post intervention with pulse oximeter to check effects of techniques applied on asthma patients.

CONTACTS AND LOCATIONS:
Overall Officials: Riffat Malik malik, Principal Investigator — Riphah International University
Locations (1):
- Sehat Medical Complex Hanjerwal, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jahan N. Effectiveness of inter costal stretch techniques among copd patients at NIDCH: Bangladesh Health Professions Institute, Faculty of Medicine, the University …; 2017.
- [Background] Trivedi D, Das AK. Effect of Intercostal Stretch and Breathing Control Exercise on Lung Function among Healthy Young Females.
- [Background] Kumar MB, Reddy RS. Immediate effect of intercostal stretch on chest expansion in healthy smokers. 2021.
- [Background] Yu L-J, Kim T-HJIJoHM, Sciences S. The effect of cervical stabilization exercises with thoracic spine extension exercises on forward head posture. 2021;9(5):852-7.
- [Background] Safarini OA, Bordoni B. Anatomy, Thorax, Ribs. 2023 Jul 10. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK538328/ PMID 30855912
- [Background] Chand, Vaish H. Effect of diaphragmatic breathing, respiratory muscle stretch gymnastics and conventional physiotherapy on chest expansion, pulmonary function and pain in patients with mechanical neck pain: A single group pretest-posttest quasi-experimental pilot study. J Bodyw Mov Ther. 2023 Oct;36:148-152. doi: 10.1016/j.jbmt.2023.07.004. Epub 2023 Jul 5. PMID 37949552
- [Background] Armstrong M, Vogiatzis I. Personalized exercise training in chronic lung diseases. Respirology. 2019 Sep;24(9):854-862. doi: 10.1111/resp.13639. Epub 2019 Jul 3. PMID 31270909
- [Background] Miller RL, Grayson MH, Strothman K. Advances in asthma: New understandings of asthma's natural history, risk factors, underlying mechanisms, and clinical management. J Allergy Clin Immunol. 2021 Dec;148(6):1430-1441. doi: 10.1016/j.jaci.2021.10.001. Epub 2021 Oct 14. PMID 34655640
- [Background] Eguiluz-Gracia I, Tay TR, Hew M, Escribese MM, Barber D, O'Hehir RE, Torres MJ. Recent developments and highlights in biomarkers in allergic diseases and asthma. Allergy. 2018 Dec;73(12):2290-2305. doi: 10.1111/all.13628. Epub 2018 Oct 30. PMID 30289997
- [Background] Osadnik CR, Gleeson C, McDonald VM, Holland AE. Pulmonary rehabilitation versus usual care for adults with asthma. Cochrane Database Syst Rev. 2022 Aug 22;8(8):CD013485. doi: 10.1002/14651858.CD013485.pub2. PMID 35993916
- [Background] Schoettler N, Strek ME. Recent Advances in Severe Asthma: From Phenotypes to Personalized Medicine. Chest. 2020 Mar;157(3):516-528. doi: 10.1016/j.chest.2019.10.009. Epub 2019 Oct 31. PMID 31678077
- [Background] Cevhertas L, Ogulur I, Maurer DJ, Burla D, Ding M, Jansen K, Koch J, Liu C, Ma S, Mitamura Y, Peng Y, Radzikowska U, Rinaldi AO, Satitsuksanoa P, Globinska A, van de Veen W, Sokolowska M, Baerenfaller K, Gao YD, Agache I, Akdis M, Akdis CA. Advances and recent developments in asthma in 2020. Allergy. 2020 Dec;75(12):3124-3146. doi: 10.1111/all.14607. Epub 2020 Oct 16. PMID 32997808
- [Background] Aaron SD, Boulet LP, Reddel HK, Gershon AS. Underdiagnosis and Overdiagnosis of Asthma. Am J Respir Crit Care Med. 2018 Oct 15;198(8):1012-1020. doi: 10.1164/rccm.201804-0682CI. PMID 29756989
- [Background] Gonzalez-Garcia M, Caballero A, Jaramillo C, Maldonado D, Torres-Duque CA. Prevalence, risk factors and underdiagnosis of asthma and wheezing in adults 40 years and older: A population-based study. J Asthma. 2015 Oct;52(8):823-30. doi: 10.3109/02770903.2015.1010733. Epub 2015 May 21. PMID 25996179
- [Background] Varraso R, Camargo CA Jr. Diet and asthma: need to account for asthma type and level of prevention. Expert Rev Respir Med. 2016 Nov;10(11):1147-1150. doi: 10.1080/17476348.2016.1240033. Epub 2016 Oct 5. No abstract available. PMID 27701925
- [Background] Sockrider M, Fussner L. What Is Asthma? Am J Respir Crit Care Med. 2020 Nov 1;202(9):P25-P26. doi: 10.1164/rccm.2029P25. No abstract available. PMID 33124914